CLINICAL TRIAL: NCT01305577
Title: Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study of ATX-101 (Sodium Deoxycholate Injection) Versus Placebo for the Reduction of Localized Subcutaneous Fat in the Submental Area
Brief Title: Evaluation of Safety and Efficacy of Deoxycholic Acid Injection (ATX-101) in the Reduction of Submental Fat
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kythera Biopharmaceuticals (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATX-101-10-16; 2010-020690-17 (EudraCT Number)
Record Dates: First submitted 2011-02-10; First posted 2011-02-28 (Estimated); Results first posted 2015-06-15 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-06

CONDITIONS: Moderate or Severe Submental Fullness
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Deoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Participants received placebo administered in 0.2 mL injections, up to 10 mL per treatment session at intervals of approximately 1 month for up to a maximum of 4 treatments.
  Interventions: Drug: Placebo
- Deoxycholic Acid Injection 1 mg/cm² (Experimental): Participants received deoxycholic acid 1 mg/cm² administered in 0.2 mL injections, up to 10 mL per treatment session at intervals of approximately 1 month for up to a maximum of 4 treatments.
  Interventions: Drug: Deoxycholic acid injection
- Deoxycholic Acid Injection 2 mg/cm² (Experimental): Participants received deoxycholic acid 2 mg/cm² administered in 0.2 mL injections, up to 10 mL per treatment session at intervals of approximately 1 month for up to a maximum of 4 treatments.
  Interventions: Drug: Deoxycholic acid injection

INTERVENTIONS:
Drug: Deoxycholic acid injection
  Other Names: ATX-101
  Arms: Deoxycholic Acid Injection 1 mg/cm²; Deoxycholic Acid Injection 2 mg/cm²
Drug: Placebo — Phosphate buffered saline placebo for injection
  Arms: Placebo

SUMMARY:
To evaluate the safety and efficacy of deoxycholic acid injection in the reduction of submental fat (fat below the chin).

ELIGIBILITY:
Inclusion Criteria:

1. Submental fat graded by the investigator as 2 or 3 using the Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) as determined on Visit 2.
2. Dissatisfaction with the submental area rated by the subject as 0, 1, 2, or 3 using the Subject Self Rating Scale (SSRS).
3. Males and nonpregnant, nonlactating females between 18 and 65 years of age, inclusive on the day of randomization. Females of childbearing potential must have a negative human chorionic gonadotropin (hCG) test result within 28 days before randomization and agree to practice medically acceptable birth control during the course of the study. Medically acceptable birth control includes: surgical sterilization, hormonal contraceptives, barrier methods or an intrauterine device (IUD).
4. History of stable body weight, in the judgment of the investigator, for at least 6 months before randomization. No significant change, in the judgment of the investigator, in diet or exercise practices for at least 6 months before randomization and agreement to not change diet or exercise practices during the course of the study.
5. Expected to comply with and understand the visit schedule and all protocol-specified tests and procedures.
6. Medically able to undergo the administration of study material determined by clinical evaluations made within 56 days before and laboratory tests obtained within 28 days before randomization for which the investigator identified no clinically significant abnormality.
7. Signed informed consent obtained before any study-specific procedure is performed.

Exclusion Criteria:

1. History of any intervention to treat submental fat (e.g., liposuction, surgery, or lipolytic agents) or trauma associated with the chin or neck areas, which in the judgment of the investigator may affect evaluation of safety or efficacy of treatment.
2. Loose skin in the neck or chin area for which reduction in submental fat may, in the judgment of the investigator, result in an aesthetically unacceptable outcome or a score of 4 on the Skin Laxity Rating Scale (SLRS).
3. Prominent platysmal bands at rest or other anatomical features that, in the judgment of the investigator, may interfere with the evaluation of submental fat or result in an aesthetically unacceptable outcome.
4. Evidence of any cause of enlargement in the submental area (e.g., thyroid enlargement or cervical adenopathy) other than localized submental fat.
5. Body mass index (BMI) greater than 30.
6. Currently on or considering starting a weight reduction regimen.
7. Any medical condition (e.g., respiratory, cardiovascular, hepatic, neurological disease, uncontrolled hypertension, or thyroid dysfunction) that would interfere with assessment of safety or efficacy or compromise the subject's ability to undergo study procedures or provide informed consent.
8. Treatment with radio frequency, laser procedures, chemical peels, or dermal fillers in the neck or chin area within 12 months before randomization, or botulinum toxin injections in the neck or chin area within 6 months before randomization.
9. History of sensitivity to any components of the study material or to topical or local anesthetics (e.g., lidocaine, benzocaine, or novocaine).
10. Previous randomization into this study or previous treatment with ATX-101.
11. Treatment with an investigational device or agent within 30 days of randomization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2010-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Beddingfield, MD, PhD, Study Director — Kythera Biopharmaceuticals, Inc.
Locations (24):
- Investigational Site, Oudenaarde, Minderbroederstaraat, Belgium
- France (5):
  - Investigational Site, Arras
  - Investigational Site, Cannes
  - Investigational Site, Nice
  - Investigational Site, Pantin
  - Investigational Site, Paris
- Germany (11):
  - Investigational Site, Augsburg
  - Investigational Site, Berlin
  - Investigational Site, Darmstadt
  - Investigational Site, Frankfurt am Main
  - Investigational Site, Landau
  - Investigational Site, Ludwigshafen
  - Investigational Site, München
  - Investigational Site, Northeim
  - Investigational Site, Potsdam
  - Investigational Site, Starnberg
  - Investigational Site, Wuppertal
- Investigational Site, Barcelona, Spain
- United Kingdom (6):
  - Investigational Site, London, London
  - Investigational Site, Salford, Manchester
  - Investigational Site, Northampton, Northampton
  - Investigational Site, Nottingham, Nottingham
  - Investigational Site, Plymouth, Plymouth
  - Investigational Site, Cheltenham

REFERENCES:
- [Derived] McDiarmid J, Ruiz JB, Lee D, Lippert S, Hartisch C, Havlickova B. Results from a pooled analysis of two European, randomized, placebo-controlled, phase 3 studies of ATX-101 for the pharmacologic reduction of excess submental fat. Aesthetic Plast Surg. 2014 Oct;38(5):849-60. doi: 10.1007/s00266-014-0364-9. Epub 2014 Jul 2. PMID 24984785

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 28 study centers in the European Union.
Pre-assignment Details: The study consisted of a 12-week treatment period and a 12-week safety follow-up period.
Period: Overall Study
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Placebo
Started | 120 | 121 | 122
Received Treatment | 119 | 121 | 122
Completed | 107 | 110 | 112
Not Completed | 13 | 11 | 10
Not completed — Adverse Event | 2 | 2 | 1
Not completed — Withdrawal by Subject | 7 | 5 | 6
Not completed — Lost to Follow-up | 4 | 3 | 2
Not completed — Protocol Deviation | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Placebo | Total
Number analyzed (Participants) | 120 | 121 | 122 | 363
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (10.94) | 46.7 (9.78) | 46.6 (10.17) | 46.4 (10.28)
Age, Customized [Number; unit: participants]
  18 - 50 years | 77 | 79 | 72 | 228
  51 - 65 years | 43 | 42 | 50 | 135
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 95 | 87 | 277
  Male | 25 | 26 | 35 | 86
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 0 | 1 | 1
  Black or African American | 2 | 2 | 0 | 4
  Hispanic or Latino | 5 | 2 | 3 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  White | 111 | 116 | 117 | 344
  Other | 1 | 1 | 1 | 3
Weight [Mean (Standard Deviation); unit: kg] | 73.83 (11.518) | 73.53 (12.413) | 73.50 (12.126) | 73.62 (11.994)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 25.94 (2.724) | 25.66 (3.063) | 25.54 (2.758) | 25.71 (2.850)
Fitzpatrick Skin Type [Number; unit: participants] — Fitzpatrick Skin Type is a numerical classification schema for human skin color and typical response to ultraviolet (UV) light:
  * Type I: Pale white skin, blue/hazel eyes, blond/red hair; Always burns, does not tan.
  * Type II: Fair skin, blue eyes; Burns easily, tans poorly.
  * Type III: Darker white skin; Tans after initial burn.
  * Type IV: Light brown skin; Burns minimally, tans easily.
  * Type V: Brown skin; Rarely burns, tans darkly easily.
  * Type VI: Dark brown or black skin; Never burns, always tans darkly.
  participants
    I-III | 108 | 109 | 99 | 316
    IV-VI | 12 | 12 | 23 | 47

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) 1-grade Response
Description: A CR-SMFRS response is defined as at least a 1-point improvement (i.e. 1-point reduction) from Baseline 12 weeks after the last treatment.
  The CR-SMFRS score is based on the investigator's clinical evaluation of the participant, where submental fullness is scored on a 5-point ordinal scale (0-4) with 0 = absent, 1 = mild, 2 = moderate, 3 = severe, and 4 = extreme.
Time Frame: Baseline and 12 weeks after last treatment (up to 24 weeks after first dose)
Population: Intent-to-treat (ITT) population, which consisted of all randomized participants who had at least one efficacy assessment (CR-SMFRS or Subject Self Rating Scale) at Baseline. Last observation carried forward (LOCF) method was used to impute missing data.
Measure: Number; unit: percentage of participants
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Placebo
Number analyzed (Participants) | 120 | 121 | 122
percentage of participants | 59.2 | 65.3 | 23.0
Statistical Analysis 1: Comparison: Deoxycholic Acid Injection 1 mg/cm² vs Placebo; The null hypothesis was there was no difference between deoxycholic acid 1 mg/cm² and placebo. An adjustment for multiplicity was performed for the two co-primary endpoints. This was accounted for by using the larger of the two P-values in the Bonferroni-Holm scheme; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Logistic regression analysis with treatment and Baseline CR-SMFRS value in the model; Odds Ratio (OR) = 4.73, 95% CI 2-sided [2.70 to 8.28] — The odds ratio was based on a logistic regression model adjusted for the Baseline score. Odds ratios >1 indicate a positive treatment effect
Statistical Analysis 2: Comparison: Deoxycholic Acid Injection 2 mg/cm² vs Placebo; The null hypothesis was there was no difference between deoxycholic acid 2 mg/cm² and placebo. An adjustment for multiplicity was performed for the two co-primary endpoints. This was accounted for by using the larger of the two P-values in the Bonferroni-Holm scheme; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Logistic regression analysis with treatment and Baseline CR-SMFRS value in the model; Odds Ratio (OR) = 6.21, 95% CI 2-sided [3.52 to 10.94] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Percentage of Participants With a CR-SMFRS 2-grade Response
Description: A CR-SMFRS 2-grade response is defined as at least a 2-point improvement (i.e. 2-point reduction) from Baseline 12 weeks after the last treatment.
  The CR-SMFRS score is based on the investigator's clinical evaluation of the participant, where submental fullness is scored on a 5-point ordinal scale (0-4) with 0 = absent, 1 = mild, 2 = moderate, 3 = severe, and 4 = extreme.
Time Frame: Baseline and 12 weeks after last treatment (up to 24 weeks after first dose)
Population: Intent-to-treat population; LOCF method was used to impute missing data
Measure: Number; unit: percentage of participants
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Placebo
Number analyzed (Participants) | 120 | 121 | 122
percentage of participants | 9.2 | 17.4 | 1.6
Statistical Analysis 1: Comparison: Deoxycholic Acid Injection 1 mg/cm² vs Placebo; Test type: Superiority or Other; p = 0.028, Regression, Logistic; Logistic regression analysis with treatment and Baseline CR-SMFRS value in the model; Odds Ratio (OR) = 5.58, 95% CI 2-sided [1.20 to 25.87] — Odds ratio was based on a logistic regression model adjusted for the Baseline score. Odds ratios >1 indicate a positive treatment effect
Statistical Analysis 2: Comparison: Deoxycholic Acid Injection 2 mg/cm² vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Logistic regression analysis with treatment and Baseline CR-SMFRS value in the model; Odds Ratio (OR) = 12.05, 95% CI 2-sided [2.75 to 52.90] — [estimate comment as in outcome 2, analysis 1]

3. Primary Outcome: Percentage of Participants With a Subject Self Rating Scale (SSRS) Response
Description: A SSRS response is defined as an SSRS score that is 4 or greater 12 weeks after the last treatment.
  The SSRS assesses participant's satisfaction with their appearance in association with the face and chin on a 7-point scale from 0 to 6: where 0 = Extremely dissatisfied, 1 = Dissatisfied, 2 = Slightly dissatisfied, 3 = Neither satisfied nor dissatisfied, 4 = Slightly satisfied, 5 = Satisfied and 6 = Extremely satisfied.
Time Frame: Baseline and 12 weeks after last treatment (up to 24 weeks after first dose)
Population: Intent-to-treat population; LOCF method was used to impute missing data
Measure: Number; unit: percentage of participants
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Placebo
Number analyzed (Participants) | 120 | 121 | 122
percentage of participants | 53.3 | 66.1 | 28.7
Statistical Analysis 1: Comparison: Deoxycholic Acid Injection 1 mg/cm² vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Logistic regression analysis with treatment and Baseline SSRS value in the model; Odds Ratio (OR) = 2.99, 95% CI 2-sided [1.74 to 5.14] — Odds ratio was based on a logistic regression model adjusted for Baseline score. Odds ratios >1 indicate a positive treatment effect
Statistical Analysis 2: Comparison: Deoxycholic Acid Injection 2 mg/cm² vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Logistic regression analysis with treatment and baseline SSRS value in the model; Odds Ratio (OR) = 5.22, 95% CI 2-sided [2.99 to 9.11] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Change From Baseline in CR-SMFRS Scores
Description: The CR-SMFRS score is based on the investigator's clinical evaluation of the participant, where submental fullness is scored on a 5-point ordinal scale (0-4) with 0 = absent, 1 = mild, 2 = moderate, 3 = severe, and 4 = extreme.
  A negative change from Baseline indicates improvement.
Time Frame: Baseline and 12 weeks after last treatment (up to 24 weeks after first dose)
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Placebo
Number analyzed (Participants) | 107 | 110 | 112
units on a scale | -0.7 (0.65) | -0.9 (0.73) | -0.2 (0.55)
Statistical Analysis 1: Comparison: Deoxycholic Acid Injection 1 mg/cm² vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Repeated Measures; The model included the fixed effect factors visit and treatment, the visit*treatment interaction, and the baseline CR-SMFRS values as covariate; LS Mean Difference = -0.51, 95% CI 2-sided [-0.68 to -0.35]
Statistical Analysis 2: Comparison: Deoxycholic Acid Injection 2 mg/cm² vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Repeated Measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.67, 95% CI 2-sided [-0.84 to -0.50]

5. Secondary Outcome: Change From Baseline in SSRS Scores
Description: The SSRS assesses participant's satisfaction with their appearance in association with the face and chin on a 7-point scale from 0 to 6: where 0 = Extremely dissatisfied, 1 = Dissatisfied, 2 = Slightly dissatisfied, 3 = Neither satisfied nor dissatisfied, 4 = Slightly satisfied, 5 = Satisfied and 6 = Extremely satisfied.
  A positive change from Baseline indicates improvement.
Time Frame: Baseline and 12 weeks after last treatment (up to 24 weeks after first dose)
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Placebo
Number analyzed (Participants) | 106 | 108 | 111
units on a scale | 2.4 (1.74) | 2.8 (1.72) | 1.4 (1.60)
Statistical Analysis 1: Comparison: Deoxycholic Acid Injection 1 mg/cm² vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; The model includes the fixed effect factor treatment and the Baseline values as covariate; LS Mean Difference = 1.04, 95% CI 2-sided [0.61 to 1.47]
Statistical Analysis 2: Comparison: Deoxycholic Acid Injection 2 mg/cm² vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; The model includes the fixed effect factor treatment and the Baseline values as covariate; LS Mean Difference = 1.41, 95% CI 2-sided [0.99 to 1.84]

6. Secondary Outcome: Change From Baseline in Submental Fat Thickness
Description: Submental thickness was measured using caliper devices.
Time Frame: Baseline and 12 weeks after last treatment (up to 24 weeks after first dose)
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Placebo
Number analyzed (Participants) | 107 | 110 | 112
mm | -3.8 (3.85) | -4.2 (3.90) | -1.7 (3.13)
Statistical Analysis 1: Comparison: Deoxycholic Acid Injection 1 mg/cm² vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Repeated Measures; The model includes the fixed effect factors visit and treatment, the visit*treatment interaction, and the Baseline values as covariate; LS mean Difference = -1.68, 95% CI 2-sided [-2.50 to -0.87]
Statistical Analysis 2: Comparison: Deoxycholic Acid Injection 2 mg/cm² vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Repeated Measures; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = -1.97, 95% CI 2-sided [-2.79 to -1.15]

7. Secondary Outcome: Change From Baseline in Patient-reported Submental Fat Rating Scale (PR-SMFRS)
Description: The PR-SMFRS is based on the participant's response to the question "How much fat do you currently have under your chin?" answered on a 5-point ordinal scale (0-4) with 0 = no chin fat at all, 1 = a slight amount of chin fat, 2 = a moderate amount of chin fat, 3 = a large amount of chin fat, and 4 = a very large amount of chin fat. Improvement is defined as any decrease in score and worsened as any increase in score.
Time Frame: Baseline and 12 weeks after last treatment (up to 24 weeks after first dose)
Population: Intent-to-treat population with available data
Measure: Number; unit: percentage of participants
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Placebo
Number analyzed (Participants) | 103 | 106 | 108
percentage of participants
  Improvement | 67.0 | 73.6 | 32.4
  No Change | 32.0 | 22.6 | 59.3
  Worsened | 1.0 | 3.8 | 8.3
Statistical Analysis 1: Comparison: Deoxycholic Acid Injection 1 mg/cm² vs Placebo; Test type: Superiority or Other; p < 0.001, Pearson's chi-square test
Statistical Analysis 2: Comparison: Deoxycholic Acid Injection 2 mg/cm² vs Placebo; Test type: Superiority or Other; p < 0.001, Pearson's chi-square test

8. Secondary Outcome: Change From Baseline in Patient-Reported Submental Fat Impact Scale (PR-SMFIS)
Description: The PR-SMFIS assesses the impact of submental fat on self-perception of 6 characteristics related to the appearance of submental fullness as evaluated by the participant. Each item is rated on an 11-point numeric scale from 0 to 10.
Time Frame: Baseline and 12 weeks after last treatment (up to 24 weeks after first dose)
Reporting Status: Not Posted, anticipated posting 2016-01

9. Secondary Outcome: Change From Baseline in Self-rating of Attractiveness
Description: Self-rating of attractiveness assesses aspects of appearance from the participant's perspective by a series of 6 questions:
  How attractive do you think your overall appearance (chin/neck, eyes, nose, mouth, entire face) is/are?" Each question was answered on a scale from 1 to 9 where 1 = Not at all attractive, 5 = Neither attractive nor unattractive and 9 = Extremely attractive.
  A positive change from Baseline indicates improvement.
Time Frame: Baseline and 12 weeks after last treatment (up to 24 weeks after first dose)
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Placebo
Number analyzed (Participants) | 101 | 104 | 105
units on a scale
  Overall Appearance | 0.9 (1.58) | 0.5 (1.44) | 0.3 (1.28)
  Chin/Neck | 1.8 (2.05) | 1.9 (2.21) | 0.5 (1.90)
  Eyes | 0.8 (1.71) | 0.1 (1.33) | 0.3 (1.27)
  Nose | 0.3 (1.34) | 0.0 (1.37) | 0.2 (1.39)
  Mouth | 0.4 (1.63) | 0.2 (1.50) | 0.3 (1.28)
  Entire Face | 0.8 (1.25) | 0.3 (1.31) | 0.0 (1.19)

10. Secondary Outcome: Change From Baseline in Derriford Appearance Scale 24 (DAS24)
Time Frame: Baseline and 12 weeks after last treatment (up to 24 weeks after first dose)
Reporting Status: Not Posted, anticipated posting 2016-01

11. Secondary Outcome: Change From Baseline in Body Image Quality of Life Inventory (BIQLI)
Time Frame: Baseline and 12 weeks after last treatment (up to 24 weeks after first dose)
Reporting Status: Not Posted, anticipated posting 2016-01

ADVERSE EVENTS:
Time Frame: From the first dose of study drug until 12 weeks after the last dose (up to 24 weeks after first treatment).
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Placebo
Serious Adverse Events (participants affected / at risk) | 1/119 | 3/121 | 2/122
Other Adverse Events (participants affected / at risk) | 111/119 | 115/121 | 75/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deoxycholic Acid Injection 1 mg/cm² (N=119) | Deoxycholic Acid Injection 2 mg/cm² (N=121) | Placebo (N=122)
Abdominal Adhesions (Gastrointestinal disorders) | 0 | 1 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Chronic Tonsillitis (Infections and infestations) | 0 | 0 | 1
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deoxycholic Acid Injection 1 mg/cm² (N=119) | Deoxycholic Acid Injection 2 mg/cm² (N=121) | Placebo (N=122)
Injection Site Pain (General disorders) | 92 | 97 | 31
Injection Site Haematoma (General disorders) | 65 | 62 | 48
Injection Site Swelling (General disorders) | 63 | 63 | 26
Injection Site Anaesthesia (General disorders) | 57 | 62 | 3
Injection Site Erythema (General disorders) | 46 | 45 | 28
Injection Site Induration (General disorders) | 22 | 33 | 3
Injection Site Oedema (General disorders) | 21 | 21 | 12
Injection Site Pruritus (General disorders) | 11 | 3 | 1
Injection Site Haemorrhage (General disorders) | 6 | 7 | 6
Injection Site Nodule (General disorders) | 1 | 9 | 0
Injection Site Warmth (General disorders) | 6 | 1 | 1
Headache (Nervous system disorders) | 8 | 7 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Study Agreement requires that the investigator or institution obtain written consent from Kythera prior to presenting and/or publishing results of this study.